CLINICAL TRIAL: NCT03857594
Title: Integrative Sequencing In Germline and Hereditary Tumours
Acronym: INSIGHT
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: INSIGHT
Record Dates: First submitted 2018-10-23; First posted 2019-02-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hereditary Cancer Syndrome; High-Risk; Mutation; Germline Mutation
Keywords: Hereditary Cancer Syndrome; High-Risk; Mutation; Germline Mutation; Rare Cancer Histology; Whole Genome Sequencing (WGS); Whole Exome Sequencing (WES)
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Archival tumor tissue, whole blood at baseline for germ-line DNA analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Individuals at risk of hereditary cancer syndrome: All individuals at risk of a hereditary cancer syndrome with or without a known germline mutation from clinical genetic testing.

SUMMARY:
This study will investigate the utility of integrative sequencing of individuals and families at risk of hereditary cancer syndromes and will uncover novel contributors to tumourigenesis. Integrative sequencing refers to:

1. Whole genome sequencing (WGS) of the germline (inherited) genome
2. Whole exome sequencing (WES) or targeted/panel sequencing of tumour(s) (somatic, tumour-specific mutations)
3. DNA methylation (methylome) analysis of tumour(s)
4. RNA sequencing (transcriptome) of tumour(s)

Eligible patients receiving genetic care at Princess Margaret Cancer Centre and the University Health Network may be approached by their genetic counsellor for participation in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥18 years of age
2. All patients and enrolled family members must have a signed and dated informed consent form

All individuals at risk of a hereditary cancer syndrome without a known germline mutation from clinical genetic testing, will be eligible for this study. This includes:

1. Individuals with multiple primary malignancies
2. Families with a strong family history of cancer suggestive of a hereditary cancer syndrome
3. Young individuals with cancer (10 years earlier than the age of onset of sporadic cases) and no identified gene mutation
4. Rare cancer histologies

Individuals with an identified germline mutation will also be eligible for this study, if there are discordant family members suggesting additional genetic factors contributing to the variable familial phenotype. For example, a family composed of mutation carriers severely affected with cancers, and carriers unaffected with cancer.

Exclusion Criteria:

None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals at risk of a hereditary cancer syndrome with or without a known germline mutation. This includes individuals with multiple primary malignancies, families with a strong family history of cancer, young individuals with cancer, rare cancer histologies.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-10-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of genomic contributors to inherited cancer through genome-wide germline analysis | Through study completion, up to 3 years
Number of identified novel mechanisms of tumorigenesis in hereditary cancer patients | Through study completion, up to 3 years

SECONDARY OUTCOMES:
Utilization rate of whole genome sequencing of the germline in identifying hereditary disorders | Through study completion, up to 3 years
Utilization rate of genome scale/targeted analysis of tumours in identifying potential therapeutic modalities | Through study completion, up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Kim, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Wang Y, Ding Q, Prokopec S, Farncombe KM, Bruce J, Casalino S, McCuaig J, Szybowska M, van Engelen K, Lerner-Ellis J, Pugh TJ, Kim RH. Germline whole genome sequencing in adults with multiple primary tumors. Fam Cancer. 2023 Oct;22(4):513-520. doi: 10.1007/s10689-023-00343-2. Epub 2023 Jul 22. PMID 37481477